CLINICAL TRIAL: NCT00475085
Title: Prevention of Delayed Nausea A Phase III Double-Blind Placebo-Controlled Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Joseph Roscoe (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Joseph Roscoe, Research Associate Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000544841; U10CA037420 (NIH); URCC-U1105 (Other: University of Rochester)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Nausea
Keywords: nausea and vomiting; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; inflammatory breast cancer; male breast cancer
MeSH Terms: conditions — Nausea; Vomiting; Breast Neoplasms; Inflammatory Breast Neoplasms; Breast Neoplasms, Male | interventions — Aprepitant; Dexamethasone; Calcium Dobesilate; Granisetron; Palonosetron; Prochlorperazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Active Comparator): Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  Interventions: Drug: dexamethasone; Drug: palonosetron hydrochloride; Drug: prochlorperazine; Drug: placebo
- Arm II (Experimental): Patients receive granisetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  Interventions: Drug: dexamethasone; Drug: granisetron hydrochloride; Drug: prochlorperazine; Drug: placebo
- Arm III (Active Comparator): Patients receive palonosetron hydrochloride IV and dexamethasone IV once on day 1, oral aprepitant once daily on days 1-3, and oral dexamethasone once daily and oral placebo twice daily on days 2 and 3.
  Interventions: Drug: aprepitant; Drug: dexamethasone; Drug: palonosetron hydrochloride; Drug: placebo
- Arm IV (Experimental): Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and oral dexamethasone once daily on days 2 and 3.
  Interventions: Drug: dexamethasone; Drug: palonosetron hydrochloride; Drug: prochlorperazine; Drug: placebo

INTERVENTIONS:
Drug: aprepitant — Given orally or IV
  Other Names: Emend
  Arms: Arm III
Drug: dexamethasone — Given orally or IV
  Other Names: Decadron
Drug: granisetron hydrochloride — Given orally or IV
  Other Names: Kytril
  Arms: Arm II
Drug: palonosetron hydrochloride — Given orally or IV
  Other Names: Aloxi
  Arms: Arm I; Arm III; Arm IV
Drug: prochlorperazine — Given orally or IV
  Other Names: Compazine
  Arms: Arm I; Arm II; Arm IV
Drug: placebo — Given orally

SUMMARY:
RATIONALE: Antiemetic drugs, such as granisetron, dexamethasone, prochlorperazine, aprepitant, and palonosetron, may help lessen or prevent nausea. It is not yet known which combination of antiemetic drugs is more effective in preventing nausea caused by chemotherapy.

PURPOSE: This randomized phase III trial is comparing different combinations of granisetron, dexamethasone, prochlorperazine, aprepitant, and palonosetron to see how well they work in preventing nausea in patients undergoing chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of palonosetron hydrochloride and dexamethasone followed by prochlorperazine with vs without dexamethasone in preventing delayed nausea in women with chemotherapy-naive breast cancer. (Arms I and IV)
* Determine if palonosetron hydrochloride is more effective than granisetron hydrochloride in controlling treatment-related delayed nausea in these patients. (Arms I and II)
* Determine if the currently recommended antiemetic guideline of aprepitant combined with palonosetron hydrochloride and dexamethasone is the most effective antiemetic regimen for controlling treatment-related delayed nausea in these patients. (Arms III and IV)

Secondary

* Determine if the addition of dexamethasone to prochlorperazine is more effective than the same regimen without dexamethasone for reducing interference with functioning caused by chemotherapy-induced nausea and vomiting in these patients. (Arms I and IV)
* Determine if palonosetron hydrochloride is more effective than granisetron hydrochloride for reducing interference with functioning caused by chemotherapy-induced nausea and vomiting in these patients. (Arms I and II)
* Determine if the currently recommended antiemetic guideline of aprepitant combined with palonosetron hydrochloride and dexamethasone is the most effective antiemetic regimen for reducing interference with functioning due to chemotherapy-induced nausea and vomiting in these patients. (Arms III and IV)

OUTLINE: This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to CCOP center and gender. Patients are randomized to 1 of 4 treatment arms. Patients receive study treatment approximately 30 minutes before their scheduled first chemotherapy treatment.

* Arm I: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
* Arm II: Patients receive granisetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
* Arm III: Patients receive palonosetron hydrochloride IV and dexamethasone IV once on day 1, oral aprepitant once daily on days 1-3, and oral dexamethasone once daily and oral placebo twice daily on days 2 and 3.
* Arm IV: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and oral dexamethasone once daily on days 2 and 3.

Quality of life is assessed at baseline and on day 4. Nausea and vomiting, fatigue, sleep quality, exercise, and the need for rescue medication (metoclopramide) are assessed on days 1-4.

PROJECTED ACCRUAL: A total of 890 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* Have a diagnosis of cancer and be chemotherapy naive.
* Must be scheduled to receive a chemotherapy treatment containing doxorubicin hydrochloride, epirubicin hydrochloride, cisplatin, carboplatin, or oxaliplatin (any dose or schedule) without concurrent radiotherapy or interferon treatment
* Chemotherapy may be for adjuvant, neoadjuvant, curative or palliative intent.
* Dose-dense regimens (e.g. chemotherapy with doxorubicin or epirubicin given every two weeks)are allowed.
* For the purposes of this study, Day 1 of chemotherapy will be defined as the day of administration of cisplatin, carboplatin, oxaliplatin, doxorubicin or epirubicin.
* Regimens with multiple-day doses of doxorubicin, epirubicin, cisplatin, carboplatin, oxaliplatin, dacarbazine, hexamethylmelamine, nitrosoureas, or streptozocin are not allowed. Chemotherapy agents, other than those listed above, may be given orally, intravenously, or by continuous infusion on one or multiple days.
* Able to understand English

Exclusion criteria:

* No symptomatic brain metastases
* No concurrent or impending bowel obstruction
* Regimens containing liposomal doxorubicin or cisplatin are not allowed.
* No concurrent pimozide, terfenadine, astemizole, or cisapride
* No concurrent doxorubicin hydrochloride liposome or cisplatin
* No concurrent multiple-day doses of dacarbazine, altretamine, nitrosoureas, streptozocin, cisplatin, carboplatin, or oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2006-12; Primary Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A. Roscoe, PhD, Principal Investigator — James P. Wilmot Cancer Center
Locations (16):
- United States (16):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhassett, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Derived] Roscoe JA, Heckler CE, Morrow GR, Mohile SG, Dakhil SR, Wade JL, Kuebler JP. Prevention of delayed nausea: a University of Rochester Cancer Center Community Clinical Oncology Program study of patients receiving chemotherapy. J Clin Oncol. 2012 Sep 20;30(27):3389-95. doi: 10.1200/JCO.2011.39.8123. Epub 2012 Aug 20. PMID 22915657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients from 15 private-practice oncology groups in the USA affiliated with the University of Rochester Cancer Center Community Clinical Oncology Program (URCC CCOP)were enrolled by research personnel from May 2007 to September 2010.
Groups:
- Arm 1 Palonosetron, Dexamethasone, Compazine: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and oral dexamethasone once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm 2 Granisetron, Dexamethasone, Compazine: Patients receive granisetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  granisetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm 3 Aprepitant, Palonosetron, Dexamethasone: Patients receive palonosetron hydrochloride IV and dexamethasone IV once on day 1, oral aprepitant once daily on days 1-3, and oral dexamethasone once daily and oral placebo twice daily on days 2 and 3.
  placebo : Given orally
  aprepitant : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm 4 Palonosetron, Dexamethasone, Compazine, Dexamethasone: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
Period: Overall Study
Arm/Group | Arm 1 Palonosetron, Dexamethasone, Compazine | Arm 2 Granisetron, Dexamethasone, Compazine | Arm 3 Aprepitant, Palonosetron, Dexamethasone | Arm 4 Palonosetron, Dexamethasone, Compazine, Dexamethasone
Started | 253 | 254 | 260 | 254
Completed | 235 | 234 | 241 | 234
Not Completed | 18 | 20 | 19 | 20

BASELINE CHARACTERISTICS:
Groups:
- Arm II: Patients receive granisetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  granisetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm III: Patients receive palonosetron hydrochloride IV and dexamethasone IV once on day 1, oral aprepitant once daily on days 1-3, and oral dexamethasone once daily and oral placebo twice daily on days 2 and 3.
  placebo : Given orally
  aprepitant : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm I: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and another oral placebo once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Arm IV: Patients receive palonosetron hydrochloride IV, dexamethasone IV, and oral placebo once on day 1 and oral prochlorperazine 3 times daily and oral dexamethasone once daily on days 2 and 3.
  placebo : Given orally
  prochlorperazine : Given orally or IV
  palonosetron hydrochloride : Given orally or IV
  dexamethasone : Given orally or IV
- Total: Total of all reporting groups
Arm/Group | Arm II | Arm III | Arm I | Arm IV | Total
Number analyzed (Participants) | 254 | 260 | 254 | 253 | 1021
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.7) | 58.6 (11.4) | 57.1 (12.4) | 58.2 (11.4) | 57.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 208 | 201 | 193 | 208 | 810
  Male | 46 | 59 | 61 | 45 | 211
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 3 | 2 | 9
  Asian | 2 | 4 | 0 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 18 | 28 | 20 | 19 | 85
  White | 232 | 226 | 231 | 229 | 918
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 254 | 260 | 254 | 253 | 1021
Previous Surgery [Number; unit: participants] | 193 | 194 | 196 | 198 | 781
Previous Radiotherapy [Number; unit: participants] | 6 | 12 | 12 | 9 | 39

OUTCOME MEASURES:

1. Primary Outcome: Home Record: Severity of Delayed Nausea
Description: 1=not at all nauseated to 7=extremely nauseated, therefore higher values are worse
Time Frame: average of day 1 afternoon, evening and night, and all of days 2 and 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm II | Arm III | Arm I | Arm IV
Number analyzed (Participants) | 234 | 241 | 234 | 235
units on a scale | 1.88 (1.27) | 1.65 (1.15) | 1.87 (1.20) | 1.68 (1.15)
Statistical Analysis 1: Comparison: Arm II vs Arm I; Group 1 - Group 2 (palonosetron vs. granisetron); Test type: Superiority or Other; p = 0.718, ANOVA — Response skewed. P-value determined after Box-Cox transformation (lambda=-1.6). Significance level set to 0.017 to account for three tested hypotheses; Testing and estimation performed using contrasts in the context of an omnibus ANOVA; Mean Difference (Final Values) = -0.013, 95% CI 2-sided [-0.225 to 0.200]
Statistical Analysis 2: Comparison: Arm I vs Arm IV; Group 1 - Group 4 (adding dexamethasone); Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 1, analysis 1]; Testing and estimation performed using contrasts in the context of an omnibus ANOVA; Mean Difference (Final Values) = 0.195, 95% CI 2-sided [-0.017 to 0.407]
Statistical Analysis 3: Comparison: Arm III vs Arm IV; Group 3 - Group 4 (aprepitant vs. prochlorperazine); Test type: Superiority or Other; p = 0.557, ANOVA — [p-value comment as in outcome 1, analysis 1]; Testing and estimation performed using contrasts in the context of an omnibus ANOVA; Mean Difference (Final Values) = -0.025, 95% CI 2-sided [-0.236 to 0.186]

ADVERSE EVENTS:
Arm/Group | Arm II | Arm III | Arm I | Arm IV
Serious Adverse Events (participants affected / at risk) | 6 | 17 | 16 | 11
Other Adverse Events (participants affected / at risk) | 1 | 1 | 0 | 1
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arm II | Arm III | Arm I | Arm IV
Lymphoma (Blood and lymphatic system disorders) | 1/254 (1) | 0/260 (0) | 0/254 (0) | 0/253 (0)
Neutropenia (Blood and lymphatic system disorders) | 0/254 (0) | 3/260 (3) | 1/254 (1) | 0/253 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Trombocytopenia (Blood and lymphatic system disorders) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Gastrointestinal (Gastrointestinal disorders) | 1/254 (1) | 3/260 (3) | 0/254 (0) | 3/253 (3)
GI Bleed (Gastrointestinal disorders) | 0/254 (0) | 0/260 (0) | 0/254 (0) | 1/253 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1/254 (1) | 1/260 (1) | 1/254 (1) | 3/253 (4)
Chest Pain (General disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 1/253 (1)
Dehydration (General disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Edema (General disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Fatigue (General disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Headache (General disorders) | 1/254 (1) | 0/260 (0) | 2/254 (2) | 0/253 (0)
Migraine (General disorders) | 0/254 (0) | 0/260 (0) | 0/254 (0) | 1/253 (2)
Restless (General disorders) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Allergic Reaction (Immune system disorders) | 0/254 (0) | 2/260 (2) | 1/254 (1) | 0/253 (0)
Infection (Infections and infestations) | 0/254 (0) | 0/260 (0) | 2/254 (2) | 0/253 (0)
MRSA (Infections and infestations) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Infusion Reaction (Injury, poisoning and procedural complications) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
Renal Failure (Renal and urinary disorders) | 1/254 (1) | 1/260 (1) | 0/254 (0) | 1/253 (1)
Hydrocele (Reproductive system and breast disorders) | 0/254 (0) | 0/260 (0) | 1/254 (1) | 0/253 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0/254 (0) | 1/260 (1) | 2/254 (2) | 0/253 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/254 (1) | 0/260 (0) | 0/254 (0) | 0/253 (0)
Hemorrhage (Vascular disorders) | 0/254 (0) | 0/260 (0) | 0/254 (0) | 1/253 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Arm II | Arm III | Arm I | Arm IV
Gastrointestinal (Gastrointestinal disorders) | 0/254 (0) | 0/260 (0) | 0/254 (0) | 1/253 (1)
Chest Pain (General disorders) | 0/254 (0) | 1/260 (1) | 0/254 (0) | 0/253 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1/254 (1) | 0/260 (0) | 0/254 (0) | 0/253 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes